CLINICAL TRIAL: NCT00456378
Title: A Prospective, Randomized, Controlled Pivotal Clinical Investigation of DIAM™ Spinal Stabilization System in Patients With Lumbar Degenerative Disc Disease.
Brief Title: Study of the Safety and Effectiveness of DIAM™ Spinal Stabilization System Versus Conservative Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision, no safety concerns
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIAM™ Device vs. Cons. Care
Record Dates: First submitted 2007-03-29; First posted 2007-04-04 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- DIAM™ spinal stabilization system (Experimental): Implantation of the DIAM Spinal Stabilization System
  Interventions: Device: DIAM™ Spinal Stabilization System
- Conservative care (Active Comparator): Conservative Care
  Interventions: Procedure: Conservative care

INTERVENTIONS:
Device: DIAM™ Spinal Stabilization System — Surgical procedure with implantation of the Investigational device
  Arms: DIAM™ spinal stabilization system
Procedure: Conservative care — Six months of conservative care, to include: patient education, medications, physical therapy and spinal injections.
  Arms: Conservative care

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of the DIAM™ Spinal Stabilization System in the treatment of moderate single-level lumbar degenerative disc disease.

DETAILED DESCRIPTION:
This pivotal clinical trial is being conducted to evaluate the DIAM™ Spinal Stabilization System for the treatment of single-level moderate lumbar degenerative disc disease. The implant under investigation in this clinical trial is the DIAM Spinal Stabilization System, and the device will be implanted using a posterior surgical approach. Patients in the control group will receive nonoperative treatment.

ELIGIBILITY:
Inclusion Criteria:

Each patient participating in this clinical trial must meet all of the following inclusion criteria:

1. Has moderate low back pain secondary to lumbar degenerative disc disease at a single level from L2 - L5. Low back pain is defined as persistent back pain, with or without radicular pain, with current episode of less than one year duration. Degenerative disc disease is confirmed by patient history, physical examination, and radiographic studies with one or more of the following factors (as measured radiographically by MRI scans or x-rays):

   * Decreased disc height >2mm, compared to the disc space at the next adjacent (superior or inferior, whichever has greater disc height) spinal level;
   * Scarring/thickening of the ligamentum flavum, annulus fibrosis, or facet joint capsule;
   * Herniated nucleus pulposus.
2. Is 18-70 years of age, inclusive, and is skeletally mature.
3. Has pre-treatment Oswestry score ≥ 30.
4. Has pre-treatment back pain score of ≥ 8 based on the Pre-Treatment Back and Leg Pain Questionnaire (Back Pain Intensity + Back Pain Frequency).
5. Has been treated nonoperatively (e.g. bed rest, physical therapy, medications, TENS, manipulation, and/or spinal injections) for a period of at least 6 weeks and not more than 6 months prior to enrollment in the clinical study.
6. If of child-bearing potential, patient is not pregnant or nursing and agrees not to become pregnant during the study period.
7. Is willing and able to participate in either of the randomized treatments for the duration of the study follow-up period. If the patient is randomized to the investigational group, he/she is willing to undergo surgery and receive the DIAM device. If the patient is randomized to the control group, he/she is willing to undergo all four nonoperative treatments.
8. Is willing and able to comply with the study plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

A patient meeting any of the following criteria is to be excluded from this clinical trial:

1. Has disc height loss > 67% at the involved level, compared to the next adjacent (superior or inferior, whichever has greater disc height) spinal level
2. Has Arachnoiditis.
3. Has a primary diagnosis of a spinal disorder other than degenerative disc disease at the involved level.
4. Requires treatment of degenerative disc disease at more than one lumbar level.
5. Has had all of the following nonoperative treatments (prescribed medications, active physical therapy, spinal injections, and patient education) within the past 6 weeks.
6. Has a sequestered herniated nucleus pulposus.
7. Has had any previous surgery at the involved or adjacent spinal levels (including procedures such as rhizotomy).
8. Has received any intradiskal ablation therapy, such as IDET.
9. Has congenital or iatrogenic posterior element insufficiency (e.g. facet resection, spondylolysis, pars fracture, or Spinal Bifida Occulta).
10. Has back pain (with or without leg, buttock, or groin pain) that is not alleviated in any spinal position.
11. Has a motor deficit of the lower extremity.
12. Has cauda equina syndrome.
13. Has compression of nerve roots with neurogenic bowel (fecal incontinence) or bladder (urinary retention or incontinence) dysfunction.
14. Has been previously diagnosed with clinically significant peripheral neuropathy.
15. Has significant vascular disease causing vascular claudication.
16. Has a medical contraindication that prevents the patient from receiving spinal injections (i.e., allergy to contrast media used to aid in placement of the needle in the epidural space).
17. Has ventral spondylolisthesis with more than 2 mm of translation at the involved level.
18. Has evidence of prior fracture or trauma to the L1, L2, L3, L4, or L5 levels in either compression or burst.
19. Has lumbar scoliosis with a Cobb angle of greater than 15°.
20. Has lumbar kyphosis or flat back syndrome.
21. Has sustained a hip fracture within the last year.
22. Has any of the following (if "Yes" to any of the below risk factors, a lumbar spine DEXA Scan will be required to determine eligibility.):

    1. Previous diagnosis of osteoporosis, osteopenia, or osteomalacia.
    2. Postmenopausal Non-Black female over 60 years of age who weighs less than 140 pounds.
    3. Postmenopausal female who has sustained a non-traumatic hip, spine or wrist fracture.
    4. Male over the age of 60 who has sustained a non-traumatic hip or spine fracture.

    If the level of DEXA T-score is -1.0 or lower (i.e., -1.5, -2.0, etc.), the patient is excluded from the study.
23. Has obesity defined by BMI greater than or equal to 40. (Refer to the BMI Table provided in the CIP.)
24. Has a documented allergy to silicone, polyethylene, titanium, or latex.
25. Has overt or active bacterial infection, either local or systemic, and/or potential for bacteremia.
26. Has a suppressed immune system or has taken steroids at any dose daily for more than one month within the last year (excluding low dose inhalers for the treatment of asthma).
27. Has a history of autoimmune disease.
28. Has presence of active malignancy or prior history of malignancy within the last 5 years (except for basal cell carcinoma of the skin).
29. Has presence or prior history of a spinal malignancy.
30. Has chronic or acute renal and/or hepatic failure or prior history of renal and/or hepatic parenchymal disease.
31. Has any disease (e.g., neuromuscular disease) that would preclude accurate clinical evaluation of the safety and effectiveness of the treatment regimens in this study.
32. Has received treatment with an investigational therapy (device and/or pharmaceutical) within 30 days prior to entering the study or such treatment is planned during the 24 months following enrollment in the study.
33. Has an implantable metal device (e.g., stimulator, pacemaker) and is unable to have an MRI.
34. Is an alcohol and/or drug abuser, as defined by currently undergoing treatment for alcohol and/or drug abuse.
35. Is mentally incompetent. If questionable, obtain psychiatric consult.
36. Has a Waddell Signs of Inorganic Behavior score of 3 or greater.
37. Is a prisoner.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2006-12; Primary Completion 2015-10-08 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Overall Success | 12 months
  A patient will be considered an overall success if all of the following conditions are met:
  1. Pain/disability (Oswestry) success;
  2. No serious adverse event classified as "implant associated", "implant-/surgical procedure associated", or "nonoperative treatment associated"; and
  3. For patients in the investigational group, no additional surgical procedure at the involved level classified as a failure. For patients in the control group, no "treatment surgery" at the involved level that was the result of a poor response to conservative care treatment.

SECONDARY OUTCOMES:
Pain/Disability Status | 12 months
  The self-administered Oswestry Low Back Pain Disability Questionnaire will be used. Success will be defined as pain/disability improvement according to the following definition:
  Pre-treatment Score - Post-treatment Score ≥ 15
Neurological Status | 12 months
  Neurological status is based on four types of measurements: motor, sensory, reflexes, and straight leg raising. Each of the sections is comprised of a number of elements. Overall neurological success will be defined as maintenance or improvement in all sections ( motor, sensory, reflex, and straightleg raising ) for the time period evaluated.
Pain Status (Back Pain and Leg Pain) | 12 months
  Numerical rating scales will be used to evaluate pain intensity and duration. The pain score (0 min, 20 Max) is derived by adding the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and duration scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Success for back pain and leg pain is described as follows: Pre-treatment Score - Post-treatment Score >0
General Health Status | 12 months
  The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) will be used to assess general health status. The SF-36 physical component summary (PCS) measures a patient's physical wellbeing and will be calculated according to algorithms formulated by the Medical Outcomes Trust. To be classified as a success, the following criterion must be met for SF-36 PCS:
  PCSPost-tx - PCSPre-tx >= 0

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Spine Institute of Arizona, Scottsdale, Arizona
  - Tower Orthopaedic & Neurosurgical Spine Institute, Beverly Hills, California
  - Los Angeles Brain and Spine Institute, Los Angeles, California
  - Neurological Surgery, Mission Viejo, California
  - Loma Linda Orthopaedic Dept, San Bernardino, California
  - Boulder Neurosurgical Associates, Boulder, Colorado
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Foundation for Orthopaedic Research and Education (FORE), Tampa, Florida
  - Georgia Neurological Surgery, Athens, Georgia
  - Dr. Sokolowski, Oak Park, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Fort Wayne Orthopaedics, Fort Wayne, Indiana
  - OrthoIndy, Indianapolis, Indiana
  - Precision Spine and Orthopaedic Specialists, Overland Park, Kansas
  - Kansas Joint & Spine Institute, Wichita, Kansas
  - Sports Medicine North Orthopaedic Surgery, Inc., Peabody, Massachusetts
  - University Physicians Group, Detroit, Michigan
  - Twin Cities Spine Center, Minneapolis, Minnesota
  - The Orthopedic Center of St. Louis, Chesterfield, Missouri
  - Advanced Neurosurgery Inc. / Kettering Medical Center, Kettering, Ohio
  - NeuroSpine Institute, Eugene, Oregon
  - Argires, Becker, Marotti, & Westphal Brain, Orthopedic/Sports Medicine & Spine Care, Lancaster, Pennsylvania
  - Orthopedic Institute, Sioux Falls, South Dakota
  - Spine Specialty Center, Memphis, Tennessee
  - Neurospine Surgical Consultants, Plano, Texas
  - Spine Team Texas, Southlake, Texas
  - The Smart Clinic, Sandy City, Utah
  - Department of Neurosurgery, University of Virginia Health System, Charlottesville, Virginia